CLINICAL TRIAL: NCT02163200
Title: Changes of Pressure on Soft Tissue Before and After Total Hip Replacement to Prevent Bedsores
Status: Withdrawn | Type: Observational
Why Stopped: due to technical issues
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Head of the Department of General Surgery, Assuta Medical Center
Other Study IDs: 0906-14
Record Dates: First submitted 2014-06-09; First posted 2014-06-13 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Transient Arthropathy of Hip
Keywords: Bedsores; pressure; hip
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pressure of total hip replacement: Patients 60 y.o. or more both sex with a history of hip arthropathy without previous bedsores or CVA

SUMMARY:
Patients candidates for total hip replacement are, generally elderlies and have hip pain, we will check if the pressure to the soft tissue changes before and after operation using a tapet with pressure sensors sending the information to specific software.

DETAILED DESCRIPTION:
one hundred Patients 60 years old and more will be considered for this study, both sexs, that have schedule for elective unilateral total hip replacement and have not bedsores previously.

All the data will be collected by FSA software, classified in an excel table. A crossover study will be performed and analyzed by a paired test.

ELIGIBILITY:
Inclusion Criteria: 60 y/o/ and more

* Both sexes
* Schedule for total hip replacement

Exclusion Criteria:

* Patient with previous bedsore
* Patients under 60 y.0.
* Previous CVA

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient 60 y.o. or more both sexs, schedule for total hip replacement, without previous bedsore
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Changes in soft tissue pressure | Day one
  Mapping of pressure will be performed twice for each patient' the first one before surgery the second one before discharge. The measure will be performed by resting, normal position

CONTACTS AND LOCATIONS:
Overall Officials: Sergio G Susmallian, MD, Study Director — Assuta MC